CLINICAL TRIAL: NCT01119131
Title: The Effects of Vitamin D on Balance in Persons With PD
Brief Title: Effects of Vitamin D in Parkinson's Disease (PD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7051-W
Record Dates: First submitted 2010-04-23; First posted 2010-05-07 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson Disease; Accidental Falls
Keywords: Vitamin D; Parkinson disease; accidental falls
MeSH Terms: conditions — Parkinson Disease | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Will be on high dose vitamin D3 (10,000 IU daily) and 1000 mg of calcium
  Interventions: Drug: Vitamin D3; Dietary Supplement: calcium
- Arm 2 (Placebo Comparator): Will be on placebo and 1000mg of calcium.
  Interventions: Dietary Supplement: calcium; Other: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 at 10,000 IU a day
  Arms: Arm 1
Dietary Supplement: calcium — 1000mg calcium daily
Other: Placebo — A placebo pill with similar appearance to the vitamin D3 will be given to those in the placebo arm
  Arms: Arm 2

SUMMARY:
A trial to measure the effects of vitamin D (versus a placebo) on balance, gait, falls, strength, and cognition in persons with Parkinson's disease.

DETAILED DESCRIPTION:
The proposed study is a randomized, double-blinded, placebo controlled intervention trial to measure the effects of vitamin D at (10,000IU/day) versus placebo on balance and falls in Parkinson's disease. The investigators will measure static, dynamic, and ambulatory balance, as well as strength, falls, and cognition before and after 16 weeks of therapy. Dynamic posturography will be used to measure static and ambulatory balance, a device called iMOBILITY will measure a timed up and go, and strength will be measured with the Biodex machine checking knee flexion and extension. Multiple quality of life and cognitive tests will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease;
* ability to ambulate 50 feet;
* ability to cooperate with balance testing;
* vitamin D level less than 40ng/ml;
* balance problems;
* ability to walk 50 feet without the help of another person

Exclusion Criteria:

* MMSE < 25;
* another neurological or orthopedic deficit that in the examiner's opinion would affect testing;
* history of renal stones or hypercalcemia;
* unwillingness to not be on other vitamin D supplementation during the study

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amie Hiller, MD BS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

REFERENCES:
- [Derived] Hiller AL, Murchison CF, Lobb BM, O'Connor S, O'Connor M, Quinn JF. A randomized, controlled pilot study of the effects of vitamin D supplementation on balance in Parkinson's disease: Does age matter? PLoS One. 2018 Sep 26;13(9):e0203637. doi: 10.1371/journal.pone.0203637. eCollection 2018. PMID 30256811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two large treatment centers in the Pacific Northwest and from the community during the time period 2011 - 2014.
Pre-assignment Details: Excluded (n=33) Not meeting criteria (n=32) (16 have vitamin D levels that were too high, 4 hx of renal stones, 3 with a history of tuberculosis, and 9 other) Lost to follow-up (n=1)
Groups:
- Vitamin D (Open Label); Vitamin D: Will be on high dose vitamin D (10,000 IU daily) and 1000 mg of calcium
  Vitamin D: Vitamin D at 10,000 IU a day
  calcium: 1000mg calcium daily
- Placebo: Will be on placebo and 1000mg of calcium.
  calcium: 1000mg calcium daily
  Placebo: A placebo pill with similar appearance to the vitamin D will be given to those in the placebo arm
Period: Overall Study
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Started | 10 | 28 | 30
Completed | 8 | 27 | 24
Not Completed | 2 | 1 | 6
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Non-Compliance | 1 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo | Total
Number analyzed (Participants) | 10 | 28 | 30 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (8.0) | 64.5 (8.0) | 68.8 (8.1) | 67.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 10 | 16
  Male | 9 | 23 | 20 | 52
Region of Enrollment [Number; unit: participants]
  United States | 10 | 28 | 30 | 68
Hoehn & Yahr [Mean (Standard Deviation); unit: units on a scale] — This is an objective staging scale for rating the clinical functioning of Parkinson's disease patients, combining functional deficits (disability) and objective signs (impairment). This staging scale is commonly used in both research settings and clinical practice. The Hoehn & Yahr is an ordinal scale ranging from 0 (no signs of disease) to 5 (wheelchair bound/bedridden). The modified version of the scale includes increments of 0.5. The HY has shown good inter-rater reliability and, although it is used worldwide, the clinimetric validity has not been established.
  units on a scale | 2.35 (0.34) | 2.48 (0.46) | 2.46 (0.47) | 2.45 (0.44)
UPDRS [Mean (Standard Deviation); unit: units on a scale] — This is the motor subsection of the UPDRS and is a commonly used tool to rate the symptoms of Parkinson's disease. Each item is rated from 0 (normal) to 4 (Can barely perform the task) several motor areas including speech, facial expression, tremor, rigidity, hand movements, agility, posture, and gait. Total score ranges from 0 to 108 with higher values on this scale represent a more severe stage of the disease.
  units on a scale | 24.20 (11.06) | 22.36 (8.56) | 25.3 (11.5) | 23.93 (10.25)
Baseline Vitamin D [Mean (Standard Deviation); unit: ng/ml] | 14.7 (3.86) | 30.21 (5.32) | 29.43 (6.46) | 27.59 (7.78)
MoCA [Mean (Standard Deviation); unit: units on a scale] — The MoCA is a short cognitive screening test designed to assist health care professionals for the detection of mild cognitive impairment. The MoCA assesses cognitive function across a variety of domains, such as visuospatial /executive functioning, naming (animals), memory, attention, language, abstraction, delayed recall, and orientation. The MoCA is scored on a 0 to 30 scale, with lower numbers indicating more cognitive impairment. A point is added to the MoCA if the subject's education high school or less (12 years or less education).
  units on a scale | 26.67 (1.94) | 24.07 (2.91) | 24.86 (3.00) | 24.78 (2.93)
Falls Self-Report [Mean (Standard Deviation); unit: Falls] | 5.86 (14.18) | 3.79 (14.85) | 3.05 (7.26) | 3.75 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Static Balance as Recorded Using Dynamic Posturography With the Sensory Organization Test (SOT 1-3)
Description: Sensory organization test (SOT) is a form of posturography. which is designed to assess quantitatively an individual's ability to use visual, proprioceptive and vestibular cues to maintain postural stability in stance. The SOT measures sway during 6 scenarios. In scenarios 1-3 the base is stable and eyes are open, then closed, and then the visual surround moves. SOT 1-3 is an average measurement of equilibrium - the average center of gravity sway for each condition. It generates a score of 0 (fall) up to 100 for each scenario and an overall composite score. Change score is measurement at 16 weeks minus measurement at baseline.
Time Frame: Baseline, 16 weeks
Population: Missing data N=2, test not performed due to participant fatigue.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 7 | 27 | 23
units on a scale | -3.25 (2.93) | 2.05 (8.85) | 1.78 (21.66)
Statistical Analysis 1: Comparison: Vitamin D (Open Label) vs Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.699, ANOVA

2. Primary Outcome: Change in Ambulatory Balance Measured by Instrumented Timed up and go (iTUG) Turn Duration
Description: This is a test that measures ambulatory balance and mobility. The instrumented timed up and go (iTUG) is an average time (seconds) of three trials that involve the participant arising from a chair, walking 25 feet turning around, walking back to the chair, and sitting down. The turn duration is the average time to turn at the end of the 25 foot walk. Longer duration of time (seconds) indicates more rigidity, a proxy measure for "ON" time in Parkinson's disease. Change score is measurement at 16 weeks minus measurement at baseline.
Time Frame: Baseline and 16 weeks
Population: Missing data N=14, test not performed due to either participant fatigue (N = 2) or mechanical/computer issues (N = 12).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 6 | 21 | 18
seconds | 0.32 (0.25) | 0.09 (0.54) | -0.07 (0.62)
Statistical Analysis 1: Comparison: Vitamin D (Open Label) vs Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.308, ANOVA

3. Primary Outcome: Change in Strength as Recorded by Measuring Knee Flexion Using Biodex (Total Work)
Description: Defined as the total muscular force output for the repetition with the greatest amount of work. The equation for work is: W = F x D. Change score is measurement at 16 weeks minus measurement at baseline.
Time Frame: Baseline, 16 weeks
Population: Missing data N=4, test not performed due to participant fatigue (N = 2), mechanical/computer issues (N = 1), illness of operator (N = 1).
Measure: Mean (Standard Deviation); unit: foot pounds
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 7 | 26 | 22
foot pounds | 83.07 (117.40) | 6.89 (176.40) | 35.19 (80.74)
Statistical Analysis 1: Comparison: Vitamin D (Open Label) vs Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.419, ANOVA

4. Secondary Outcome: Change in Cognition (Trail Making Test B-A)
Description: The Trail Making Test (TMT) consists of two parts (A & B) in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test provides information about visual search speed, scanning, speed of processing, and executive functioning. Part A measures processing speed and part B measures executive functioning. The TMT is time to complete each part of the test in seconds. Higher scores indicate greater impairment. Subtracting part A from part B is theorized to reduce the influence of the working memory and visuospatial demands and, therefore, provides a relatively pure indicator of executive function. Change score is measurement (Part B - Part A) at 16 weeks minus measurement (Part B - Part A) at baseline, negative scores indicate a improvement in executive functioning.
Time Frame: Baseline, 16 weeks
Population: Missing data (N = 8) due to scheduling difficulties (N = 3), neuropsychological administration errors (N = 2), patient discontinuing (N = 1), maximum time allowance met and discontinued test (N = 2).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 7 | 23 | 21
seconds | 8.00 (30.89) | 12.13 (49.83) | -17.33 (74.7)
Statistical Analysis 1: Comparison: Vitamin D (Open Label) vs Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.253, ANOVA

5. Secondary Outcome: Change in Quality of Life as Recorded Using Quality of Life Scales (PDQ39)
Description: The PDQ39 is a 39 item patient completed survey targeting well-being and functioning in PD. This scale address 8 dimensions (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort). The PDQ39 dimension scores are on a scale of 0 ("Never") to 4 ("Always/Cannot Do"). Scale scores are summed and range from 0 to 100 with 100 being the maximum level of problems. For a single index figure to characterize the impact of Parkinson's disease upon PD patients (PDSI), all 39 items of the PDQ39 can be summed. The PDQ39 and the use of a PDSI have shown adequate reliability and convergent validity. Change score is measurement at 16 weeks minus baseline measurement, negative scores indicate an improvement in quality of life.
Time Frame: Baseline, 16 weeks
Population: Missing data (N = 3), patient forgot form and did not return mailed form (N = 3).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 8 | 24 | 24
units on a scale | -0.16 (0.96) | -0.02 (0.47) | -0.14 (0.79)
Statistical Analysis 1: Comparison: Vitamin D (Open Label) vs Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.793, ANOVA

6. Primary Outcome: Change in Dynamic Balance as Recorded Using Dynamic Posturography With the Sensory Organization Test (SOT 4-6)
Description: Sensory organization test (SOT) is a form of posturography. which is designed to assess quantitatively an individual's ability to use visual, proprioceptive and vestibular cues to maintain postural stability in stance. The SOT measures sway during 6 scenarios. In 4-6 the base moves and the subject has eyes open, then closed, then the visual surround moves. SOT 4-6 is an average measurement of equilibrium - the average center of gravity sway for each condition. It generates a score of 0 (fall) up to 100 for each scenario and an overall composite score. Change score is measurement at 16 weeks minus measurement at baseline.
Time Frame: Baseline, 16 weeks
Population: Missing data N=3, test not performed due to participant fatigue (N = 2) or computer/mechanical error (N = 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 7 | 27 | 22
units on a scale | -1.56 (11.91) | 2.272 (12.63) | -1.89 (14.23)

7. Primary Outcome: Change in Strength as Recorded by Measuring Knee Extension Using Biodex (Total Work)
Description: as for outcome 3
Time Frame: Baseline, 16 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: foot pounds
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 7 | 26 | 22
foot pounds | 18.11 (66.65) | 23.33 (83.16) | 17.49 (32.02)
Statistical Analysis 1: Comparison: Vitamin D (Open Label) vs Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.949, ANOVA

8. Secondary Outcome: Change in Parkinsonism as Measured by the UPDRS
Description: This is the motor subsection of the UPDRS and is a commonly used tool to rate the symptoms of Parkinson's disease. This scale rates from 0 (normal) to 4 (Can barely perform the task) several motor areas including speech, facial expression, tremor, rigidity, hand movements, agility, posture, and gait. A sum score represents motor function with higher values on this scale represent a more severe stage of the disease. Change is measurement at 16 weeks minus baseline measurement, negative scores indicate an improvement in Parkinson's motor symptoms.
Time Frame: Baseline, 16 weeks
Population: Missing data (N = 2), invalid sum due to missing rating (N = 1), not completed due to scheduling conflicts (N = 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Number analyzed (Participants) | 8 | 27 | 22
units on a scale | 0.25 (8.33) | 0.48 (5.60) | -0.18 (9.73)
Statistical Analysis 1: Comparison: Vitamin D (Open Label) vs Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.957, ANOVA

ADVERSE EVENTS:
Arm/Group | Vitamin D (Open Label) | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 1/10 | 1/28 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (Open Label) (N=10) | Vitamin D (N=28) | Placebo (N=30)
Illness (General disorders) | 1 (1) | 1 (1) | 1 (1) — Non-Specified Illness
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes